CLINICAL TRIAL: NCT04891172
Title: Phase II/III Clinical Trial Study to Evaluate Efficacy and Safety of Anti COVID 19 Intravenous Immunoglobulin (C-IVIG) Therapy for Severe COVID-19 Patients
Brief Title: Anti COVID 19 Hyperimmune Intravenous Immunoglobulin (C-IVIG) Therapy for Severe COVID-19 Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Collaborators: Higher Education Commission (Pakistan) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-IVIG-02
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: COVID19 (Corona Virus Disease-2019); SARS-CoV-2 (Severe Acute respiratory syndrome Coronavirus 2); Passive immunization; Intravenous Immunoglobulin (IVIG); Pooled Convalescent Plasma; Severe ill COVID-19 patients; Antibody; Anti COVID 19 Antibodies; Anti SARS CoV 2 Antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The Control group will be receive Standard of care only
- C-IVIG (Experimental): The intervention group will receive the single dose of C-IVIG (0.15g/kg) with Standard of Care
  Interventions: Biological: Anti COVID 19 Intravenous Immunoglobulin (C-IVIG)

INTERVENTIONS:
Biological: Anti COVID 19 Intravenous Immunoglobulin (C-IVIG) — Intervention arm will receive single dose of 0.15g/kg C-IVIG. This will be infused within period of 16 hours intravenously. Additionally, all participants will receive same standard care.
  Standard Care as per hospital protocol, which may include:
  Airway support, Anti-Viral medication, Antibiotics, Fluid Resuscitation, Hemodynamic Support, Steroids, Painkillers, Anti-Pyretics, anti coagulant
  Arms: C-IVIG

SUMMARY:
Severe ill Patients will be enrolled in the study (n=310) after duly filled consent forms. Recipients will be divided into 2 group, each group contain 155 patients to compare Safety and efficacy of patients in Clinical Trial phase II/III. One Group will receive 0.15g/kg single dose of anti COVID 19 intravenously immunoglobulin (C-IVIG) develop from convalescent plasma of recovered patients from COVID 19, along with Standard of care. The Comparator group will only receive standard of Care

DETAILED DESCRIPTION:
The research team at Dow University of Health Sciences has purified immunoglobulin (both SARS-CoV 2 antibodies and existing antibodies) from convalescent plasma of COVID19 individuals and pooled it to prepare IVIG formulation to treat severe and critically ill COVID-19 patients. Phase I/II trial was completed and showed potential safety and efficacy of the drug Anti COVID-19 intravenous immunoglobulin (C-IVIG) in severe and critical patients with COVID-19.

This trial's aim is to investigate the safety and efficacy of passive immunization in severe COVID-19 patients in phase II/III. The trial will be a randomized, single-blinded, superiority trial, through parallel-group design. The participant will either receive C-IVIG with Standard of care or receive only Standard of care. The study will consist of 310 participants of which 155 will receive a single dose of C-IVIG (0.15g/kg) with the standard of care and 155 will receive only the standard of care. Standard of care is standard hospital care which includes airway support, anti-viral medication, antibiotics, fluid resuscitation, hemodynamic support, steroids, painkillers, and antipyretics.

Randomized test patients will receive a single dose of C-IVIG in the following two dosage groups:

Group 1 (Test): Severe COVID-19 patients: Single dose of 0.15g/Kg with standard hospital care

Group 2 (Comparator): Severe COVID-19 patients: only standard hospital care only

ELIGIBILITY:
Inclusion Criteria:

1. Above 18 years of age
2. Have positive COVID PCR on nasopharyngeal and/or oropharyngeal swabs
3. classified as severe* COVID-19 according to WHO guideline (5L-15L of oxygen requirement on FM, NRM)
4. Consent given by the patient or first degree relative

Exclusion Criteria:

1. Critical COVID-19 patients [ non-invasive ventilation (HFNC, BiPAP, CPAP) and invasive ventilation],
2. Pregnant females
3. Previous allergic reaction to immunoglobulin treatment
4. Known case of any autoimmune disorder
5. Chronic kidney disease
6. Known case of thromboembolic disorder
7. Aseptic meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-02 (Estimated)

PRIMARY OUTCOMES:
28 day Mortality | 28 days
  All cause mortality of participants will be monitored for 28 days to asses the safety and efficacy of C-IVIG

SECONDARY OUTCOMES:
Immediate and serious adverse event during hospital Stay | 28 days
  Immediate adverse event (within 24 hours) and serious adverse event (throughout the hospital stay) which will be observed
Clinical Status of follow-up days according to 7-Catergory Ordinal Scale | 28 days
  Clinical Status of follow-up days according to 7-Catergory Ordinal Scale
  1. Not hospitalized and no limitations of activities
  2. Not hospitalized, with limitation of activities, home oxygen requirement, or both
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring any supplemental oxygen
  5. Hospitalized, requiring noninvasive ventilation or use of high-flow oxygen devices
  6. Hospitalized, receiving invasive mechanical ventilation
  7. Death
change in C-Reactive Protein (CRP) levels | 5 Days
  Change in C-Reactive protein (CRP) levels form enrollment (baseline) till 3 days followup to monitor inflammation
change in interleukin 6 (IL-6) | 5 days
  Change in IL-6 levels form enrollment (baseline) till 3 days followup
change in anti-SARS-CoV-2 antibody levels | 5 days
  Change in IL-6 levels form enrollment (baseline) till 3 days followup by quantitive method
change in Horowitz idex | 28 days
  The Horowitz index is a ratio used to assess lung function in patients during Hospital stay
change in radiological findings | 5 days
  Change in any radiological after receive single Dose of C-IVIG

CONTACTS AND LOCATIONS:
Overall Officials: Shaukat Ali, PhD, Principal Investigator — Dow University of Health Sciences, Principal Dow College of Biotechnology
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Ali S, Luxmi S, Anjum F, Muhaymin SM, Uddin SM, Ali A, Ali MR, Tauheed S, Khan M, Bajwa M, Baig SU, Shalim E, Ahmed I, Khan AS, Quraishy S. Hyperimmune anti-COVID-19 IVIG (C-IVIG) Therapy for Passive Immunization of Severe and Critically Ill COVID-19 Patients: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Nov 2;21(1):905. doi: 10.1186/s13063-020-04839-5. PMID 33138867
- [Background] Ali S, Uddin SM, Ali A, Anjum F, Ali R, Shalim E, Khan M, Ahmed I, M Muhaymin S, Bukhari U, Luxmi S, Khan AS, Quraishy S. Production of hyperimmune anti-SARS-CoV-2 intravenous immunoglobulin from pooled COVID-19 convalescent plasma. Immunotherapy. 2021 Apr;13(5):397-407. doi: 10.2217/imt-2020-0263. Epub 2021 Feb 9. PMID 33557591
- [Background] Xie Y, Cao S, Dong H, Li Q, Chen E, Zhang W, Yang L, Fu S, Wang R. Effect of regular intravenous immunoglobulin therapy on prognosis of severe pneumonia in patients with COVID-19. J Infect. 2020 Aug;81(2):318-356. doi: 10.1016/j.jinf.2020.03.044. Epub 2020 Apr 10. No abstract available. PMID 32283154
- [Background] Chai KL, Valk SJ, Piechotta V, Kimber C, Monsef I, Doree C, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Oct 12;10:CD013600. doi: 10.1002/14651858.CD013600.pub3. PMID 33044747
- [Derived] Kimber C, Valk SJ, Chai KL, Piechotta V, Iannizzi C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Hyperimmune immunoglobulin for people with COVID-19. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD015167. doi: 10.1002/14651858.CD015167.pub2. PMID 36700518
- [Derived] Ali S, Shalim E, Farhan F, Anjum F, Ali A, Uddin SM, Shahab F, Haider M, Ahmed I, Ali MR, Khan S, Rao S, Guriro K, Elahi S, Ali M, Mushtaq T, Sayeed MA, Muhaymin SM, Luxmi S, Saifullah, Qureshi S. Phase II/III trial of hyperimmune anti-COVID-19 intravenous immunoglobulin (C-IVIG) therapy in severe COVID-19 patients: study protocol for a randomized controlled trial. Trials. 2022 Nov 8;23(1):932. doi: 10.1186/s13063-022-06860-2. PMID 36348476

DOCUMENTS (1):
  • Study Protocol: Protocol00 (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT04891172/Prot_001.pdf